CLINICAL TRIAL: NCT03915509
Title: Evaluation Of The Effect Of Surface Properties On The Stabılıty Of The Different Implants With Resonance Frequency Analysis
Brief Title: Evaluation Of The Effect Of Surface Properties On The Stabılıty Of The Different Implants
Acronym: Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Burcu Gürsoytrak, Assistant Proffesor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2011-31
Record Dates: First submitted 2019-04-05; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Dental Implantation
Keywords: nanotopography; osseointegration; resonance frequency analysis.
MeSH Terms: interventions — Resonance Frequency Analysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive group (Experimental): In this study different surfaced implants applied patients who has bilateral edentulous mandibular molar region In one hemiarch, an alkali-modified surfaced implants were applied (bioactive group); in the other hemiarch, sand-blasted surfaced implants were applied (sand-blasted group). The implants were randomly selected.
  Interventions: Device: Evaluation of the effect of surface properties on the stability of the different implants with resonance frequency analysis
- Sandblasted group (Active Comparator): In this study different surfaced implants applied patients who has bilateral edentulous mandibular molar region In one hemiarch, an alkali-modified surfaced implants were applied (bioactive group); in the other hemiarch, sand-blasted surfaced implants were applied (sand-blasted group). The implants were randomly selected.
  Interventions: Device: Evaluation of the effect of surface properties on the stability of the different implants with resonance frequency analysis

INTERVENTIONS:
Device: Evaluation of the effect of surface properties on the stability of the different implants with resonance frequency analysis — Lasak Impladent Implants (sandblasted)
  Other Names: Lasak Impladent Implants (hydrophilic surface)

SUMMARY:
This randomised clinical study aims to evaluate different surfaced implants (alkali-modified surfaced implants or sand-blasted surfaced implants) stability with resonance frequency analysis(RFA).

DETAILED DESCRIPTION:
This is randomised controlled double blind study. Fourteen patients (8 women and 6 men;age 43.7 ± 8.56 years) who were attending the Oral and Maxillofacial Surgery Department and scheduled for implant placement surgery were included in this study. Dental implants were placed using one-stage protocol. After adminstration of local anesthesia (Ultracain DS; Aventis Pharmaceuticals, Istanbul, Turkey ), an incision was made on the alveolar ridge. A total of 50 implants (Impladent implants from the Lasak) were placed in the not site assignement mandibular premolar/molar sites according to the manufacturer's instructions. To prevent bias which implant to the right or left to make the decision investigators decided by envelope. The person making the measurement does not know which surface implant is made to the patient. An equal number of implants were applied simultaneously with different surfaces. The patient does not know where the implant is placed. All used implants were 3.7 width, 10mm. height and same design for standardization this study. Investigators obtained good primarly stability and placed a healing cap for 45 implants . 3 sandblasted and acid-and alkali-treated surface straight (bioactive)implants and 2 sandblasted surface straight implants were excluded in this study for bad primary stability. Investigators used to measure implant stability with Osstell ISQ ( Integration diagnostic AB, Savedalen, Sweden) for each implant at the time of surgery before flap closure, 2. week,6. week and 12. week postoperatively.This device was used in both buccolingual and mesiodistal direction. The Smartpegs (Integration Diagnostics AB, Göteborg, Sweden) were compressed and the measurements were performed by the same surgeon for standardization of the stability measurements. The measurements were taken twice in the buccolingual direction and twice in the mesiodistal direction. The arithmetic mean of the 2 measurements from each direction was regarded as the representative ISQ of that implant. In addition, each implant was clinically evaluated at all visits for mobility, pain, and signs of infection.

ELIGIBILITY:
Inclusion Criteria:

1.A healthy medical condition (ASA 1 and ASA 2 according to the American Society of Anesthesiologists classification) 2.The ability to withstand the stress of dental implant surgery 3.The need for bilateral implant-supported rehabilitation in the mandibular premolar/molar area.

-

Exclusion Criteria:

1. An active infection or severe inflammation in the areas intended for implant placement
2. Metabolic bone disorder
3. Uncontrolled diabetes
4. Hematologic disorder
5. Need for bone augmentation
6. The smokers
7. Drug users (anti-inflammatory agents, bisphosphonates)
8. Pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Survey | 3 months
  Defined after clinical and radiological examination.

SECONDARY OUTCOMES:
Surgery Implant Stability Quotient Measurement | 3 months
  After insertion of the implant, the primary stability measured implant stability quotient at the end of implantation with resonance frequency analysis.The implant stability quotient (range: 0-100) is a conversion of the resonance frequency value (3,500 to 8,500 Hz) . Generally, implant stability quotient values are interpreted as follows: i) >70: high stability, ii) 60-69: medium stability, and iii) <60: low stability.
Second Implant Stability Quotient Measurement | 3 months
  After insertion of the implant, the primary stability measured implant stability quotient after two weeks later.The implant stability quotient (range: 0-100) is a implantation with resonance frequency analysis.The implant stability quotient (range: 0-100) is a conversion of the resonance frequency value (3,500 to 8,500 Hz) . Generally, implant stability quotient values are interpreted as follows: i) >70: high stability, ii) 60-69: medium stability, and iii) <60: low stability.
Third Implant Stability Quotient Measurement | 3 months
  After insertion of the implant, the primary stability measured implant stability quotient after six weeks later.The implant stability quotient (range: 0-100) is a implantation with resonance frequency analysis.The implant stability quotient (range: 0-100) is a conversion of the resonance frequency value (3,500 to 8,500 Hz) . Generally, implant stability quotient values are interpreted as follows: i) >70: high stability, ii) 60-69: medium stability, and iii) <60: low stability.
Fourth Implant Stability Quotient Measurement | 3 months
  After insertion of the implant, the primary stability measured ISQ after twelve weeks later.The ISQ (range: 0-100) is a implantation with resonance frequency analysis.The ISQ (range: 0-100) is a conversion of the resonance frequency value (3,500 to 8,500 Hz) . Generally, ISQ values are interpreted as follows: i) >70: high stability, ii) 60-69: medium stability, and iii) <60: low stability.

CONTACTS AND LOCATIONS:
Overall Officials: Hanife ATAOGLU, Proffesor, Study Director — Selcuk University
Locations (1):
- Aydın Adnan Menderes University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anil S, Al Dosari A. Impact of bone quality and implant type on the primary stability: an experimental study using bovine bone. J Oral Implantol. 2015;41:144-148. Balshi T.J., Wolfinger G.J.: Immediate loading of Branemark implants in edentulous mandibles: a preliminary report. Implant Dentistry., 1997; 6:83-8. Barewal R M, Oates T W, Meredith N, Cochran D L. Resonance frequency measurement of implant stability in vivo on implants with a sandblasted and acid-etched surface. Int J Oral Maxillofac İmplants, 2003; 18,:641-651. Bischof M, Nedir R, Szmukler-Moncler S, Bernard J P, Samson J. Implant stability measurement of delayed and immediatelly loaded implants during healing . A clinical RFA study with SLA ITI ımplants. Clin Oral Implants Res 2004;15: 529-539. Branemark PI. Introduction to osseointegration. In:Branemark PI, Zarb GA, Albrektsson T, eds. Tissue-Integrated Prostheses in Osseointegration in Clinical Dentistry. Chicago: Quintessence Pub Co Inc; 1985: 11-14. Cameron HU, Pilliar RM, Mac Nab I. The effect of movement on the bonding of porous metal to bone. J Biomed Mater Res. 1973;7:301-311. Cochran DL., Buser D. Bone response to sandblasted and acid-attacked titanium: Experimental and clinical studies In: Davies J E. Bone Engineering. Toronto: Em Squared; 2000:391-398. Davies JE. Mechanism of endosseous integration. Int J Prosthodont, 1998; 11: 391-401.